CLINICAL TRIAL: NCT06986993
Title: Impact of Semaglutide Administration on Tobacco Use Behavior and Related Mechanisms Among Smokers With Obesity
Brief Title: Impact of Semaglutide on Tobacco Use and Related Health Behaviors
Acronym: ONSET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ONSET
Record Dates: First submitted 2025-05-13; First posted 2025-05-23 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — semaglutide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a double blind randomized placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blind to the intervention condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Active Comparator): Participants will be randomized to receive active semaglutide or placebo (saline) injection once a week for 12weeks
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will be randomized to receive active semaglutide or placebo (saline) injection once a week for 12weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Participants are randomized to receive either semaglutide or placebo (saline) via sc injection once a week for 12 weeks. Dose will be titrated per recommendations every 4 weeks,starting at .25mg, then 0.5mg and then 1.0mg
  Other Names: Ozempic
  Arms: Semaglutide
Drug: Placebo — Participants are randomized to receive either semaglutide or placebo (saline) via sc injection once a week for 12 weeks. Dose will be titrated per recommendations every 4 weeks,starting at .25mg, then 0.5mg and then 1.0mg
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This pilot randomized trial will assess the impact of 12 weeks of semaglutide administration (vs placebo) on changes in: (i) tobacco use and related factors (nicotine craving, withdrawal, motivation to quit, etc.) and (ii) biological biomarkers of health (e.g., epigenetics, glucose variability via continuous glucose monitoring [CGM], etc.) in adult smokers with obesity (n = 40). We will integrate molecular biology procedures (e.g., epigenetics) to maximize internal validity with real-world smartphone-based ecological momentary assessment (EMA) surveys to maximize external validity

ELIGIBILITY:
Inclusion criteria :

1. Aged 18-65;
2. report daily use of >2 cigarettes per day (CPD), as this is a sufficient threshold for detecting tobacco use disorder, per MPI Oliver's published work57;
3. meet criteria for obesity (BMI ≥30 kg/m2); and
4. no immediate desire to quit tobacco use (using criteria form the clinical practice guidelines for treating tobacco dependence)

Exclusion criteria:

1. Severe psychiatric disturbance precluding successful completion of the study, defined as

   a. Ever schizophrenia, schizoaffective disorder, or bipolar disorder (assessed at the screener and again at baseline); b. Psychiatric hospitalization in the past year (assessed at the screener and again at baseline); c. Suicidal ideation in the past month or any past year suicide attempt (assessed at baseline) i. Suicidal ideation determined by the Ask Suicide Screening Questions (ASQ) Question 1-3 ii. Any suicide attempts in the past year (ASQ 4) iii. Suicidal intent and plan (ASQ 5) iv. PHQ-9 score of 20 or higher, indicating severe depression or PHQ-9 score of 15 or higher if participant also indicates worsening of symptoms in the past 3 months.

   v. Worsening symptoms of depression or anxiety in the past 3-months (as determined by Medical History Questionnaire).
2. personal or family history of medullary thyroid carcinoma, multiple endocrine neoplasia syndrome, and personal history of pancreatitis, type I or type II diabetes, diabetic retinopathy, or gastroparesis;
3. current use of nicotine replacement therapy or other quit smoking medication;
4. history of bariatric surgery;
5. Current or past 6-month use of a GLP-1 agonist or any other weight-lowering/anti-obesity or glucose-lowering medications. These include (but are not limited to: sulfonylurea, insulin, metformin, thiazolidinediones (TZD), dipeptidyl peptidase-4 (DPP-IV) inhibitors, sodium-glucose cotransporter-2 (SGLT-2) inhibitors, or GLP-1 analogs.
6. Clinical labs out of range/unacceptable:

   1. creatinine ≥ 2 mg/dL, eGFR ≤ 60 mL/min/1.73 m2,
   2. triglycerides> 500 mg/dl,
   3. ALP > 4x the upper normal limit,
   4. abnormal blood lipase levels,
   5. other substantially abnormal clinical lab values as determined by the Study Practitioner
   6. A1C 6.5% or higher
   7. Glucose >126 mL fasting or >200mg/dL random
   8. Alanine aminotransferase (ALT) >3x upper normal limit
7. History of significant gastrointestinal disorder, including inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if in remission), diverticular disease, severe gastroparesis, diagnosis of mega-rectum or colon, congenital anorectal malformation, or clinically significant rectocele, intestinal or colonic obstruction, or suspected intestinal obstruction, intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), pancreatitis, active biliary disease
8. Any other reason or clinical condition that the investigators judge would interfere with study participation and/or be unsafe for a possible subject.
9. Known or suspected allergy to semaglutide, any of the product components, or any other GLP-1 analogue.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Cigarette smoking | 12 weeks
  Changes in number of cigarettes smoked per day

SECONDARY OUTCOMES:
Weight | 12 weeks
  change in weight (in lbs)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
This is a small-scale feasibility study with very limited resources to manage data sharing and support efforts by other investigators.